CLINICAL TRIAL: NCT06251921
Title: The Chromatic Evaluation of Universal Nano-hybrid Composites
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Prodan Corina Mirela, Dr., Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1032/55
Record Dates: First submitted 2024-01-28; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Healthy Lifestyle
Keywords: resin-based composite; color; pre-heated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restorations 1 (Experimental): preheated resin-based composite
  Interventions: Procedure: Restoration
- Restorations 2 (Experimental): room temperature resin-based composite
  Interventions: Procedure: Restoration

INTERVENTIONS:
Procedure: Restoration — with resin-based composite

SUMMARY:
The goal of this clinical trial is to evaluate the preheating effect of a group shade resin-based composite. The evaluation will be done on Ryge criteria. The main question it aims to answer is if there is a difference in time between preheated and non-heated resin-based composites in the oral cavity. Participants will be given treatment for cavities class 2 on premolars and molar and will come for recall at 24h, 1 week, 6 weeks, 3 months, 6 months, and 1 year.

DETAILED DESCRIPTION:
The participants in the study will be adult patients (over 18 years old). Each patient will receive 2 restorations on premolars or molars, class 2, and medium cavities. The restorations will be performed under isolation with rubber-dam, and restored with preheated or not-heated resin-based composite. The occlusion will be tested and they will be notified to come for recall in order to make the evaluation of the restorations.

ELIGIBILITY:
Inclusion Criteria:

* Permanent dentition
* The OHI index = 0
* Non-smoking patient
* The patient has a healthy diet
* The patient has parafunction
* The antagonist tooth is healthy / with direct restorations
* The caries are situated on proximal surfaces on premolars, molars
* The cavities have a medium depth

Exclusion Criteria:

* Temporary dentition
* The OHI index >= 1
* The patient is smoker
* The patient has an unhealthy diet
* The patient suffers from bruxism, clenching
* The antagonist tooth has an indirect restoration
* The caries are situated on canines or incisors
* The cavities have a deep or shallow depth

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Clinical inspection of the restorations | 24 hours
  The blind observer will clinically inspect the restorations , following the Ryge scale criteria
Clinical inspection of the restorations | 1 week
  The blind observer will clinically inspect the restorations , following the Ryge scale criteria
Clinical inspection of the restorations | 6 weeks
  The blind observer will clinically inspect the restorations , following the Ryge scale criteria
Clinical inspection of the restorations | 1 year
  The blind observer will clinically inspect the restorations , following the Ryge scale criteria

CONTACTS AND LOCATIONS:
Overall Officials: Diana Dudea, DDS, Study Director — Iuliu Hațeganu University of Medicine and Pharmacy
Locations (1):
- GlobalDent, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: Yes
The data collected will be used to publish in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year after the data is collected
Access Criteria: the data will be provided to the statistician